CLINICAL TRIAL: NCT01108133
Title: Neural and Pharmacological Correlates of Intrusions in Patients With Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GC-fMRI-PTSD; GC-fMRI-PTSD-2010 (Other: Intern)
Record Dates: First submitted 2010-04-20; First posted 2010-04-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2016-07

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; Traumatic Memories; fMRI
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hydrocortisone, fMRI, Intrusions (Experimental): 10 mg Hydrocortisone are administered one hour before the fMRI experiment. We use the script-driven imagery paradigm to induce intrusive memories during fMRI scanning.
  Interventions: Drug: 10 mg HydrocortisoneHöchst
- Dexamethasone, fMRI, Intrusions (Experimental): 2 mg Dexamethasone are administered at 10 pm the day before the fMRI experiment. (DEX-Test). We use the script-driven imaging paradigm to induce intrusive memories during fMRI-scanning.
  Interventions: Drug: Dexamethasone
- Placebo, fMRI, Intrusions (Experimental): Placebo is administered one hour before the fMRI experiment. We use the script-driven imaging paradigm to induce intrusive memories during fMRI-scanning in patients with posttraumatic stress disorder.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 10 mg HydrocortisoneHöchst — 10 mg Hydrocortisone Höchst are administered one hour before fMRI scanning
  Other Names: HydrocortisoneHöchst
  Arms: Hydrocortisone, fMRI, Intrusions
Drug: Dexamethasone — 2 mg Dexamethasone are administered at 10 pm the day before the fMRI experiment.
  Arms: Dexamethasone, fMRI, Intrusions
Drug: Placebo — Placebo
  Arms: Placebo, fMRI, Intrusions

SUMMARY:
There is evidence that glucocorticoids have an impact on intrusive memories in patients with posttraumatic stress disorder (PTSD). Hydrocortisone impairs intrusive memory retrieval whereas dexamethasone should strengthen intrusions in PTSD. We, the investigators, want to investigate (1) the effect of these two glucocorticoids on traumatic memories and (2) assess the neural correlates using the script-driven imagery paradigm in the functional magnetic resonance imaging (fMRI) scanner. We hypothesize that intrusive memories are less intensive under hydrocortisone-administration and more intense under dexamethasone-administration comparing both to a placebo-condition. Regarding the neural activation pattern we expect higher activation in the hydrocortisone condition in the amygdala, the hippocampus and the medial prefrontal cortex compared to the placebo-condition and less activation in the dexamethasone-condition compared to the placebo-condition.

DETAILED DESCRIPTION:
There is evidence that glucocorticoids have an impact on intrusive memories in patients with posttraumatic stress disorder (PTSD). Hydrocortisone impairs intrusive memory retrieval whereas dexamethasone should strengthen intrusions in PTSD. We, the investigators, want to investigate (1) the effect of these two glucocorticoids on traumatic memories and (2) assess the neural correlates using the script-driven imagery paradigm in the functional magnetic resonance imaging (fMRI) scanner. Therefore an individual trauma-and an individual neutral -script is assessed from each participant, recorded and replayed during fMRI-scanning. We hypothesize that intrusive memories are less intense under hydrocortisone-administration and more intense under dexamethasone-administration comparing both to a placebo-condition. Regarding the neural activation pattern we expect higher activation in the hydrocortisone condition in the amygdala, the hippocampus and the medial prefrontal cortex compared to the placebo-condition and less activation in the dexamethasone-condition compared to the placebo-condition.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45
* Female
* Posttraumatic Stress Disorder assessed by the Structured Clinical Interview (SKID-I)
* Intrusive memories (Impact of Events Scale - Revised [IES-R] intrusion scale > 7)

Exclusion Criteria:

* • Lifetime diagnosis schizophrenia according to Diagnostic and Statistical Manual, Fourth Edition (DSM-IV)

  * Mental retardation
  * Body mass index < 16.5
  * Current drug and alcohol abuse and addiction
  * Life-threatening self-injurious behavior in the last 4 months
  * Suicide attempt with the strong intention to die in the last 4 months.
  * Following diseases in anamnesis: stomach ulcera or intestinal ulcera, pancreatitis, corticoid-induced psychosis, severe osteoporosis, severe hyper-tension, heart failure, myasthenia gravis, asthma bronchiale, glaucoma, cataract, diabetes mellitus, herpes simples, herpes zoster (viremic phase), renal transplantation.
  * Any pretreatment with hydrocortisone in the last 4 weeks prior to the first administration of Investigational Medicinal Product.
  * Following current medication: cardiac glycosides, saluretics, antidiabetics, cumarin-derivatives, rifampicine, phenytoine, barbiturates, primidone, non-steroidal anti-inflammatory drug (NSAID), salicylate and indometacine, atropine, praziquantel, chloroquine, hydroxychloroquine, mefloquine, somatropine, protireline, cyclosporine, non-depolarising muscle relaxants.
  * Pregnancy or lactation period
  * Inadequate birth control
  * Shift working
  * Intercontinental travel within 2 weeks prior to enrollment (to avoid jet-lag)
  * History of hypersensitivity to investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product.
  * No subject will be allowed to enrol in this trial more than once.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Neural activation pattern of intrusive memories in patients with posttraumatic stress disorder under administration of hydrocortisone, dexamethasone and placebo. | May 2010-Sept 2011

SECONDARY OUTCOMES:
Intensity of intrusions under the administration of hydrocortisone, dexamethasone and placebo. | may 2010-Sept. 2011

CONTACTS AND LOCATIONS:
Overall Officials: Christian Schmahl, MD, Principal Investigator — Central Institute of Mental Health, Dep. of Psychosomatic and Psychotherapeutic Medicine
Locations (1):
- Central Institute of Mental Health, Dep. of Psychosomatic and Psychotherapeutic Medicine, Mannheim, Baden Württemberg6, Germany

IPD SHARING:
Plan to Share IPD: No